CLINICAL TRIAL: NCT05874232
Title: The Impact of Heartfulness Self-Care Program on Anxiety, Satisfaction With Life, and Loneliness Levels in Students and Staff in High Schools.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heartfulness Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022/01/2
Record Dates: First submitted 2023-04-04; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Satisfaction With Life; Loneliness
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heartfulness Group (Experimental): Participants were asked to practice relaxation tools for 15 minutes a day using the calendar and HeartBot app, and participate in once a weekly webinar for 30 minutes during the four weeks. The GAD, SWLS, and UCLA Loneliness scale was recorded prior to the start of the study, at the end of the program at Week 4, and after the duration of 4 weeks at Week 8. The score was reviewed to see the changes in anxiety, satisfaction with life, and loneliness scale.
  Interventions: Behavioral: Self-Care Program through Heartfulness
- Control Group (No Intervention): The control group had no change in their daily routines.

INTERVENTIONS:
Behavioral: Self-Care Program through Heartfulness — A four-week Self-Care program through Heartfulness will be offered to participants in the Heartfulness group. This would include a daily practice of relaxation tools for 15 minutes a day using an app and once a weekly webinar for 30 minutes. Guided relaxation and meditation sessions will be offered to the participants during the intervention weeks. These virtual sessions were conducted by Heartfulness Champions and certified trainers from Heartfulness Institute.
  Arms: Heartfulness Group

SUMMARY:
This quantitative study assesses the baseline anxiety, satisfaction with life, and loneliness scores in students and staff in a global study. Assessments at baseline will include the GAD, SWLS, and UCLA loneliness scale, and the same questionnaires were collected in Week 4 and Week 8. The Google form questionnaire will ask the high schoolers and staff for their email address and their parent's email address (if they are under 18). The form will also include a question eliciting interest in participation in the 4-weeks Heartfulness program. The program will include tools that promote a heart-based nurturing environment focusing on relaxation, positivity, and developing growth mindsets.

DETAILED DESCRIPTION:
The specific aim of this study is to assess changes in scores measuring symptoms of anxiety using GAD-7 (and GAD-Child), Satisfaction with Life Scale (SWLS and SWLS-C), and UCLA Loneliness Scale (Version 3).

ELIGIBILITY:
Inclusion Criteria:

* High School Students (grades 9-12) and Staff, aged 14 and above, and willing to participate in the study.

Exclusion Criteria:

* Non-English speaking high school students and staff and those with mental health diagnoses such as Major Depressive Disorder and Anxiety disorders.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-07-03 (Actual)

PRIMARY OUTCOMES:
Assess the current level of Anxiety | Week 0
  To assess the current level of anxiety in high school students and staff through GAD Scale.
Changes level of Anxiety | Week 4 and Week 8
  To assess the beneficial impact of Heartfulness program on anxiety in high school students and staff.
Assess the current level of Satisfaction with Life | Week 0
  To assess the current level of satisfaction with life in high school students and staff through SWLS Scale.
Changes level of Satisfaction with Life | Week 4 and Week 8
  To assess the beneficial impact of Heartfulness program on satisfaction with life in high school students and staff.
Assess the current level of Loneliness | Week 0
  To assess the current level of loneliness in high school students and staff through UCLA loneliness scale.
Changes in Loneliness levels | Week 4 and Week 8
  To assess the beneficial impact of Heartfulness program on loneliness in high school students and staff.

CONTACTS AND LOCATIONS:
Locations (1):
- Ranjani B Iyer, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Publish a research paper with details on the study design, protocol, analysis of data, and report on implications to stress management and wellness tools.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting six months after publication
Access Criteria: Access criteria IPD and any additional supporting information will be shared with the researchers furthering research in stress management and emotional wellness tools.

REFERENCES:
- [Derived] Iyer P, Iyer L, Carter N, Iyer R, Stirling A, Priya L, Sriraman U. Self-Care Program as a Tool for Alleviating Anxiety and Loneliness and Promoting Satisfaction With Life in High School Students and Staff: Randomized Survey Study. JMIR Form Res. 2024 Sep 30;8:e56355. doi: 10.2196/56355. PMID 39047180